CLINICAL TRIAL: NCT03236311
Title: A Randomized, Double-blind, Placebo-controlled Parallel Arm Dose Titration Study to Assess the Effects of SAR407899 in Patients With Microvascular Angina (MVA) and/or Persistent Stable Angina Despite Angiographically Successful Percutaneous Coronary Intervention (PCI)
Brief Title: A Dose Titration Study to Assess the Effects of SAR407899 in Patients With MVA and/or Persistent Stable Angina Despite Angiographically Successful PCI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: (Recruitment was early terminated due to slow recruitment. Not linked to any safety concern.)
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT14656; 2016-000629-38; U1111-1182-1709 (Other: UTN)
Record Dates: First submitted 2017-07-24; First posted 2017-08-01 (Actual); Results first posted 2019-07-11 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Microvascular Coronary Artery Disease
MeSH Terms: interventions — Adenosine; regadenoson

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo for 4 weeks.
  Interventions: Drug: Placebo; Drug: Adenosine; Drug: Regadenoson; Drug: 13N-ammonia; Drug: 82Rubidium
- SAR407899 (Experimental): SAR407899 with dose titration over 4 weeks administration (3 week titration phase + 1 week maintenance phase).
  Interventions: Drug: SAR407899; Drug: Adenosine; Drug: Regadenoson; Drug: 13N-ammonia; Drug: 82Rubidium

INTERVENTIONS:
Drug: SAR407899 — Pharmaceutical form: Capsule Route of administration: Oral
  Arms: SAR407899
Drug: Placebo — Pharmaceutical form: Capsule Route of administration: Oral
  Arms: Placebo
Drug: Adenosine — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Regadenoson — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: 13N-ammonia — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: 82Rubidium — Pharmaceutical form: Solution for injection Route of administration: Intravenous

SUMMARY:
Primary Objective:

To assess the effects of SAR407899 on coronary vasomotor function using the coronary flow reserve (CFR) in participants with microvascular angina (MVA) and/or persistent stable angina despite angiographically successful percutaneous coronary intervention (PCI).

Secondary Objectives:

* To assess the effects of SAR407899 on quality of life using Seattle Angina Questionnaire physical limitation scale (SAQ-PL) in participants with MVA and/or persistent stable angina despite angiographically successful PCI.
* To assess the safety of SAR407899 in participants with MVA and/or persistent stable angina despite angiographically successful PCI with a focus on identified risks such as hypotension and orthostatic hypotension.
* To assess SAR407899 plasma concentrations in MVA participants and/or persistent stable angina despite angiographically successful PCI.

DETAILED DESCRIPTION:
The total duration of study per participant was:

- up to 9 weeks for participants with previous coronary artery angiography or coronary computed tomography angiography (CCTA) within 24 months prior to screening with up to 4 weeks screening period, 3 weeks titration phase, 1 week maintenance period, and 1 week follow-up after the last investigational medicinal product administration.

or

- up to 11 weeks for participants with previous coronary artery angiography or CCTA between 24 months and 5 years prior to screening who need CCTA during screening period with up to 6 weeks screening period, 3 weeks titration phase, 1 week maintenance period, and 1 week follow-up after the last investigational medicinal product administration.

ELIGIBILITY:
Inclusion criteria:

* Male or female participants not at childbearing potential >=18 year-old or legal age of majority.
* Female participant if she has undergone sterilization at least 3 months earlier or was post-menopausal.
* Post-menopausal status was defined by having no menses for 12 months without an alternative medical cause.
* In females not treated with hormonal replacement therapy (HRT), menopausal status was confirmed by a high follicle stimulating hormone (FSH) level greater than 40 international units per litre (IU/L).
* In females on HRT and whose menopausal status was in doubt (i.e. in women aged less than 45 years), a highly effective contraception methods was required. Contraception was used during the whole study and for at least seven days corresponding to time needed to eliminate study treatment.
* Symptomatic stable angina pectoris (typical or atypical symptoms with an average of at least bi-weekly episodes over the past month).
* Participants with non-obstructive (<50% stenosis) coronary arteries or intermediate stenosis (between 50 and 70%) should have fractional flow reserve (FFR) >0.80 or instantaneous wave-free ratio (iFR) >0.89 on angiogram, documented within the previous 24 months*. In participants with stenting, a minimum diameter stenosis of <10% is required.

or Coronary computed tomography angiography (CCTA) with finding of non-obstructive coronary arteries within the past 24 months* in participants without previous percutaneous coronary intervention (PCI).

*Note: in cases of clinically suspected progression of atherosclerosis as per the Investigator, a more contemporary (i.e., 6 months) evidence should be provided.

or CCTA performed during screening period, with finding of non-obstructive coronary arteries, in participants diagnosed with microvascular angina (MVA) and stable angina without previous PCI who did not have a coronary angiogram or CCTA in the previous 24 months but between 24 months to 5 years.

- Baseline global coronary flow reserve (CFR) (measured during the study) assessed by 13N-ammonia or 82Rubidium positron emission tomography (PET) scan <2.0.

Exclusion criteria:

* Any use of nitrates (except short-acting nitrates) and/or dipyridamole and/or phosphodiesterase type 5 (PDE 5) inhibitors within one week prior to baseline PET scan or anticipated to be used during the study.
* Esophageal dysmotility or esophagitis.
* Participants with acute coronary syndrome (ACS) (myocardial infarction [MI] and/or unstable angina) in previous 3 months.
* Unsuccessful or incomplete coronary revascularization with residual obstructive stenosis or coronary artery disease (CAD) progression in native vessels as documented on invasive coronary angiography (>=50% stenosis) within 24 months of enrollment.
* Percutaneous coronary intervention performed at the time of an ACS (MI or unstable angina) in the previous 12 months.
* Recent PCI within the past 3 months.
* Participants with history of coronary artery bypass grafting (CABG).
* Recent (<=3 months) major surgery (i.e. valvular surgery, surgery for congenital heart disease), stroke, transient ischemic attack [TIA], sustained ventricular arrhythmia, clinically significant structural heart disease (moderate-severe valvular disease, hypertrophic cardiomyopathy, congenital heart disease, pulmonary hypertension).
* Regional local flow abnormal perfusion defects at baseline PET scan*.

  *Note: if contemporary evidence with invasive coronary angiography or CCTA demonstrates non-obstructive coronary arteries or if the regional local flow abnormal perfusion defect on PET scan is consistent with previous studies then participant qualifies for the study.
* Participants with cardiac conduction abnormalities (second or third degree atrioventricular [AV] block, sick sinus syndrome, symptomatic bradycardia, sinus node disease) except in participants fitted with a functioning pacemaker.
* History or known carotid stenosis:
* Carotid stenosis (>50%) or
* History of carotid stenosis in participants with previous symptoms.
* Contraindication or known hypersensitivity to adenosine or regadenoson.
* Contraindication to aminophylline.
* Contraindication to vasodilator stress PET scan and/or CCTA if CCTA needed during screening.
* Inability to discontinue treatment with methylxanthines treatment within 24 hours prior to PET scan.
* Participant unable to read, understand and fill a questionnaire without any help (eg, partially visually impaired or blind).
* Systolic blood pressure (SBP) <110 millimeter of mercury (mmHg) at baseline.
* Presence at baseline of symptomatic orthostatic hypotension (SBP decrease of 20 mmHg or more at Minute 3 or Minute 5 between seated and standing position), or asymptomatic orthostatic hypotension with a decrease in SBP equal or greater than 30 mmHg at Minute 3 or Minute 5 when changing from the seated to the standing position.
* Renal impairment with estimated glomerular filtration rate (eGFR) <50 milliliter/minute/1.73 square meter (mL/min/1.73 m^2) at screening and baseline.
* Drug-induced liver injury related criteria:
* Underlying hepatobiliary disease.
* Alanine Aminotransferase (ALT) >3 times the upper limit of normal (ULN).

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- United States (6):
  - Investigational Site Number 8400003, Los Angeles, California
  - Investigational Site Number 8400001, Jacksonville, Florida
  - Investigational Site Number 8400013, Wellington, Florida
  - Investigational Site Number 8400008, Baltimore, Maryland
  - Investigational Site Number 8400006, Boston, Massachusetts
  - Investigational Site Number 8400010, Philadelphia, Pennsylvania
- Investigational Site Number 2080001, København NV, Denmark
- Investigational Site Number 5280001, Nijmegen, Netherlands
- Investigational Site Number 4100002, Seoul, South Korea
- Investigational Site Number 7520001, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in United States, South Korea, Sweden, Netherlands and Denmark from 12 Oct 2017 to 23 Jul 2018.
Pre-assignment Details: A total of 10 participants who met all of the inclusion criteria and none of the exclusion criteria were randomized and enrolled in the study.
Period: Overall Study
Arm/Group | Placebo | SAR407899
Started | 5 | 5
Completed | 5 | 2
Not Completed | 0 | 3
Not completed — Study terminated by sponsor | 0 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Randomized population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SAR407899 | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.3) | 57.2 (8.5) | 61.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Uncorrected Global Coronary Flow Reserve (CFR) at Week 4
Description: Absolute change from baseline to Week 4 in uncorrected global CFR, as assessed by the central core laboratory. The global CFR is the ratio of absolute myocardial blood flow (MBF) at stress over that at rest. The MBF was assessed by 13N-ammonia or 82Rubidium positron emission tomography (PET) scan.
Time Frame: Baseline, Week 4
Population: Analysis was performed on modified intent-to-treat (mITT) population that included all randomized participants analyzed according to the treatment group allocated by randomization; who received at least 1 dose or part of a dose of the investigational medicinal product (IMP) and with an evaluable primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | SAR407899
Number analyzed (Participants) | 4 | 2
ratio | 0.5 (0.6) | 0.2 (0.7)

2. Secondary Outcome: Change From Baseline in Angina-induced Physical Limitation Assessed Using Seattle Angina Questionnaire Physical Limitation Scale (SAQ-PL) at Week 4
Description: The SAQ-PL measures how common daily activities representing low, medium, and high exertional requirements were limited by angina (9 items). It was scored by assigning each response an ordinal value, beginning with 1 for the response that implied the 'lowest level of functioning' to 5 for 'not at all limited', and summing across the 9 items. The score of 9 items was then transformed to 0-100 range by subtracting the lowest possible scale score, dividing by the range of the scale and multiplying by 100. The range of scores was 0 to 100, with higher scores indicates better functioning. A change of 10 points was considered to be clinically important.
Time Frame: Baseline, Week 4
Population: As the number of participants randomized fell well below target (10 vs. 78), hence no data was collected and no analysis was performed.
Arm/Group | Placebo | SAR407899
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pharmacokinetic Parameter: SAR407899 Plasma Concentration
Time Frame: Day 1, 8, 15, 22, and Day 29
Population: as for outcome 2
Arm/Group | Placebo | SAR407899
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from signature of the informed consent form up to the end of follow up (up to Week 5 post-treatment follow-up visit)
Description: Reported AEs are treatment-emergent adverse events that is AEs that developed/worsened during 'the treatment emergent period' (the time from the first dose of study drug administration up to 7 days after the last dose of study drug administration). Analysis was performed on the safety population which included all randomized participants who received at least one dose or part of a dose of the IMP.
Arm/Group | Placebo | SAR407899
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | SAR407899 (N=5)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sports Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (5)
Dizziness Postural (Nervous system disorders) | 0 (0) | 1 (4)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to small number of participants entering randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT03236311/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT03236311/SAP_001.pdf